CLINICAL TRIAL: NCT02657980
Title: The Effect of tDCS in Patients With Moderate to Severe Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ybrain Inc. (Industry)
Collaborators: Severance Hospital (Other); Gangnam Severance Hospital (Other); Myongji Hospital (Other); CHA University (Other); National Health Insurance Service Ilsan Hospital (Other); Ajou University (Other); Hallym University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUL003MDD
Record Dates: First submitted 2015-06-22; First posted 2016-01-18 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; tDCS; MDD; transcranial Direct Current Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YBand(YDT-201N) (Experimental): transcranial Direct Current Stimulation (tDCS) application 5 days a week for 2 weeks (total of 10 applications)
  Interventions: Device: Yband(YDT-201N)
- Sham-Yband(YDT-201N) (Sham Comparator): sham-tDCS application 5 days a week for 2 weeks (total of 10 applications)
  Interventions: Device: Sham-Yband(YDT-201N)

INTERVENTIONS:
Device: Yband(YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 30 min; 30 sec of ramp-up and -down; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: YBand(YDT-201N)
Device: Sham-Yband(YDT-201N) — transcranial Direct Current Stimulation (tDCS) 2mA for 30 sec; left (anode) and right (cathode) Dorsolateral prefrontal cortex (DLPFC)
  Arms: Sham-Yband(YDT-201N)

SUMMARY:
Study Type: Interventional Study Design: Allocation: Randomized Endpoint Classification: Safety/Efficacy Study Intervention Model: Parallel Assignment Masking: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor) Primary Purpose: Treatment

DETAILED DESCRIPTION:
Patients will be randomized to receive either real or sham-tDCS as well as anti-depressant drugs. tDCS will be applied over the left (anode) and right (cathode) dorsolateral prefrontal cortex (DLPFC). Patients will visit the hospital to get tDCS administrations 5 days a week for 2 weeks. They will be evaluated every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of a major depressive disorder as confirmed by the SCID-IV and MINI (without psychotic features)
* Greater than 22 points of Montgomery-Asberg Depression Rating Scale
* Aged 19 to 65.
* Has provided informed consent

Exclusion Criteria:

* Has other mental disorders diagnosed by Axis-I, except major depressive disorder (However, subject who is diagnosed as both major depressive disorder as well as anxiety disorder can participate the study.)
* History of suicidal attempt in the last 6 months
* Diagnosed with bipolar or psychotic major depressive disorder
* Diagnosed with other depressive disorders: dysthymic disorder, and depressive disorders that are not elsewhere classified.
* Has hypersensitivity to sertraline ingredients
* A score of 5 or greater for the question #10 in MADRS
* Diagnosed with closed angle glaucoma or has a history of glaucoma.
* History of participation in other clinical trials within 30days.
* A major and/or unstable medical or neurologic illness
* Currently taking substances that contain sertraline, mono amine oxidase inhibitor, or pimozide
* Pregnant or has a positive pregnancy serum test.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms as assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | from baseline to Week 6
  Measured by Montgomery-Åsberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Effect of tDCS on Depressive Symptoms as assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | At 6 weeks after treatment.
  The percentage of subjects whose MADRS score decreases over 50% against the base in week 6 after treatment.
Effect of tDCS on questionnaire results as assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) | At 6 weeks after treatment
  The percentage of subjects whose MADRS score is under 10 in week 6 after treatment.
Average change in results for 2, 4, 6 weeks after treatment as assessed by the clinician-rated Clinical Global Impression-Severity of Illness Scale (CGISI) | At 2 weeks, 4 weeks and 6 weeks after treatment
  Average change of CGISI at 2 weeks, 4 weeks and 6 weeks after treatment compare to the base respectively.
Average change in results for 2, 4, 6 weeks after treatment as assessed by Korean-Beck Depression Inventory-II (K-BDI-II) | At 2 weeks, 4 weeks and 6 weeks after treatment
  Average change of K-BDI-II at 2 weeks, 4 weeks and 6 weeks after treatment compare to the base respectively.
Average change in results for 2, 4, 6 weeks after treatment as assessed by Korean-Beck Anxiety Depression Inventory (K-BAI) | At 2 weeks, 4 weeks and 6 weeks after treatment
  Average change of K-BAI at 2 weeks, 4 weeks and 6 weeks after treatment compare to the base respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Seungwoo Lee, Study Director — Ybrain Company
Locations (1):
- Ybrain, Seoul, South Korea